CLINICAL TRIAL: NCT03673267
Title: Nutricity: A Pilot Study to Improve Parental Nutrition Literacy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 142565
Record Dates: First submitted 2018-08-28; First posted 2018-09-17 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Dietary Habits; Dietary Modification; Literacy; Knowledge, Attitudes, Practice
Keywords: health literacy; nutrition literacy; parenting
MeSH Terms: conditions — Feeding Behavior; Literacy; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutricity (Experimental)
  Interventions: Behavioral: Nutricity

INTERVENTIONS:
Behavioral: Nutricity — Participants will use their smartphone or web-accessing device to access the Nutricity website to potentially increase nutrition literacy and set nutrition goals. Participants will have their own user name and password to access the site. Access to Nutricity will last approximately 3 months.

SUMMARY:
The aim of this study is to engage parents and their young children (1-5 years of age) using the mobile intervention, Nutricity. Study goals are to increase parental nutrition literacy and improve eating habits of children.

DETAILED DESCRIPTION:
Nutricity website: Nutricity is a mobile website that uses communication techniques that break down each section to teach parents and children the nutrition information. The site addresses five components of nutrition literacy:

1. ability to comprehend nutrition text
2. eating foods in the right portions
3. using food labels to make nutrition decisions
4. grouping foods into like categories
5. choosing between similar foods (consumer skills)

Participants will have three months of free access to Nutricity during this study. They will also be encouraged to set one nutrition goal per week and encouraged to use Nutricity to help attain that goal. Participants will send weekly goals through text message to a number provided by the research team.

There are three phases to this study:

Baseline: Participants will be asked to come to the clinic or research lab 1 time for procedures and assessments that will help the investigator assess nutrition literacy and eligibility.

Nutricity: During this phase participants will use their smartphone to access the Nutricity website to potentially increase nutrition literacy and set nutrition goals.

This phase will last approximately 3 months.

End Study: Participants will be asked to come to the research lab 1 time to perform the same procedures and assessments completed in the baseline visit.

Assessments include:

Height/Weight: Parent/guardian and child will have their height and weight measured.

Demographics: questionnaires will ask for information such as name, date of birth and race.

Nutrition Questionnaires: Participants will complete 1 questionnaire on 2 occasions to assess nutrition literacy using the Nutrition Literacy Assessment Instrument (NLit). The NLit measures nutrition literacy and is comprised of six domains:

1. nutrition and health
2. energy sources in food
3. household food measurement
4. food labels/numbers
5. food groups
6. consumer skills

Parents/Guardians will also be asked about fruit, vegetable, fat, and fiber intake.

24-hour Recall: Parents will be asked questions about a child's current diet over the previous 24 hours. For children who eat meals at school or daycare, researchers will provide forms to the child's teacher or daycare provider to record the meals they eat while there. Two additional recalls will be done during the study that will be done with researchers over the phone.

Resonance Raman Spectroscopy (Veggie Meter): During this assessment, the veggie meter will apply gentle pressure to the pad of a child's fingertip to put it in close contact with light, to detect and measure carotenoid in the blood. Carotenoids are the yellow, orange, and red colors that are produced in plants, such as tomatoes. Three, 10-45 second measurements are taken and averaged for the recorded score.

Exit Survey: Upon completion of the study, participants will complete one questionnaire to provide the researchers feedback on their experience in the study.

ELIGIBILITY:
Inclusion Criteria:

* Parents must be English speaking and must 1) Identify as primary food decision-maker for the home, 2) Have internet access at home and 3) Must have a device for accessing the internet. Smartphones, owned by ~75-92% of the target population, are adequate to satisfy the latter two criteria.

Exclusion Criteria:

* 1) Overt cognitive or psychiatric illness, 2) Visual impairments that preclude reading survey instruments or using a tablet, 3) Child illness requiring a highly restrictive diet, such as renal disease, celiac disease, etc., 4) Planning to travel internationally during the study, 5) child is a foster child or ward of the state.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2019-08-12 (Actual)

PRIMARY OUTCOMES:
Parental Nutrition Literacy | 12 weeks
  Measured by the Nutrition Literacy Assessment Instrument

SECONDARY OUTCOMES:
Child Diet Quality | 12 weeks
  Measured by Healthy Eating Index derived from 3 24 hour recalls obtained at baseline and end of study

OTHER OUTCOMES:
Skin Carotenoid Content | 12 weeks
  Resonance Raman spectroscopy ("Veggie Meter," Longevity Link Corporation) uses gentle pressure applied to the pad of the fingertip to put in close contact with light to detect and measure carotenoid molecules in the blood. Three, 10-45 second measurements are taken and averaged for the recorded score.

CONTACTS AND LOCATIONS:
Overall Officials: Heather D Gibbs, PhD, RD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: Undecided